CLINICAL TRIAL: NCT02335255
Title: A Multi-Center, Double-Blind, Randomized, Parallel-Group, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Naftifine Hydrochloride Gel 2% and Naftin® (Naftifine Hydrochloride) Gel 2% in Patients With Tinea Pedis.
Brief Title: Evaluate Safety and Efficacy of Naftifine Hydrochloride Gel 2% and Naftin® Gel 2% in Tinea Pedis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NFTC 1409-1722
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Tinea Pedis
MeSH Terms: conditions — Tinea Pedis | interventions — naftifine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Naftifine Hydrochloride Gel 2% (Experimental): Naftifine Hydrochloride Gel 2% (Taro Pharmaceuticals Inc.)
  Interventions: Drug: Naftifine Hydrochloride Gel 2%
- Naftin® Gel 2% (Active Comparator): Naftin® (Naftifine Hydrochloride) Gel 2% (Merz Pharmaceuticals, LLC)
  Interventions: Drug: Naftin® Gel 2%
- Placebo Topical Gel (Placebo Comparator): Placebo Topical Gel (Taro Pharmaceuticals Inc.)
  Interventions: Drug: Placebo Topical Gel

INTERVENTIONS:
Drug: Naftifine Hydrochloride Gel 2% — Naftifine Hydrochloride Gel 2% applied once daily for fourteen consecutive days to affected areas plus a 1/2 inch margin of healthy surrounding skin.
  Other Names: Naftifine
  Arms: Naftifine Hydrochloride Gel 2%
Drug: Naftin® Gel 2% — Naftin® Gel 2% applied once daily for fourteen consecutive days to affected areas plus a 1/2 inch margin of healthy surrounding skin.
  Other Names: Naftifine
  Arms: Naftin® Gel 2%
Drug: Placebo Topical Gel — Placebo Topical Gel applied once daily for fourteen consecutive days to affected areas plus a 1/2 inch margin of healthy surrounding skin.
  Other Names: Vehicle
  Arms: Placebo Topical Gel

SUMMARY:
To compare the efficacy and safety of the test formulation Naftifine Hydrochloride Gel 2% to Naftin® (Naftifine Hydrochloride) Gel 2%

DETAILED DESCRIPTION:
The purpose of this study is to compare the efficacy and safety of the test formulation Naftifine Hydrochloride Gel 2% to Naftin® (Naftifine Hydrochloride) Gel 2% in a six week study (four weeks after the end of two week treatment) in patients with tinea pedis.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating females 18 years of age or older.
* The sum of the clinical signs and symptoms scores of the target lesion is at least 4, including a minimum score of at least 2 for erythema and a minimum score of 2 for either scaling or pruritus.
* Clinical diagnosis of interdigital tinea pedis with lesions localized to the interdigital spaces or predominantly interdigital, but may extend to other areas of the foot.
* The presence of interdigital tinea pedis infection, confirmed by the observation of segmented fungal hyphae during a microscopic potassium hydroxide wet mount preparation.

Exclusion Criteria:

* Females who are pregnant, lactating or planning to become pregnant during the study period.
* Use of antipruritics, including antihistamines within 72 hours prior to baseline visit.
* Use of topical corticosteroids, antibiotics or antifungal therapies within 2 weeks prior to baseline visit.
* Use of systemic corticosteroids, antibiotics or antifungal therapies within 1 month prior to baseline visit.
* Use of oral Terbinafine or Itraconazole within 2 months prior to baseline visit.
* Use of immunosuppressive medication or radiation therapy within 3 months prior to baseline visit.
* Any known hypersensitivity to Naftifine Hydrochloride, or any component of the formulation.
* Confluent, diffuse moccasin-type tinea pedis of the entire plantar surface.
* History of significant or current evidence of chronic infectious disease, system disorder, organ disorder, or other medical condition that would place patient at undue risk by participation or could jeopardize the integrity of the study evaluations.
* Evidence of any concurrent dermatophytic infection of the toe nails or dermatological condition of the foot that may interfere with the investigator's evaluation of tinea pedis.
* Patients with a past history of dermatophyte infections with a lack of response to antifungal therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1519 (Actual)
Dates: Start 2014-06-27 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Therapeutic cure after end of treatment | Study day 38-46
  The proportion of subjects with therapeutic cure, defined as both mycological cure and clinical cure, at the test-of-cure visit conducted four weeks after the end of treatment (study day 38-46).

CONTACTS AND LOCATIONS:
Overall Officials: Catawba Research, Study Chair — http://catawbaresearch.com/contact/

IPD SHARING:
Plan to Share IPD: No